CLINICAL TRIAL: NCT03848052
Title: Epidemiological Strategy and Medical Economic (ESME) Research Program / Academic Real World Data Platform: Evolution of the Therapeutic Care in Lung Cancer in France Since 2015
Brief Title: Evolution of the Therapeutic Care in Lung Cancer in France Since 2015 (ESME LC)
Status: Recruiting | Type: Observational
Sponsor: UNICANCER (Other)
Collaborators: AstraZeneca (Industry); Merck Sharp & Dohme LLC (Industry); Roche Pharma AG (Industry); Pfizer (Industry); Bristol-Myers Squibb (Industry); Janssen, LP (Industry); Amgen (Industry); Daiichi Sankyo (Industry); Pierre Fabre Medicament (Industry); QUINTEN HEALTH (Unknown)
Responsible Party: Sponsor
Other Study IDs: ESME LC
Record Dates: First submitted 2018-01-25; First posted 2019-02-20 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-12

CONDITIONS: Lung Cancer
Keywords: lung cancer; observational study; survival; real world data; real life setting
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This database compiles data from existing data available from patient's electronic medical records (EMR) at the 38 participating hospitals (20 French comprehensive cancer centers and 18 public hospitals).

DETAILED DESCRIPTION:
The database includes data related to patient demographics, tumor characteristics (diagnosis, histology, relapses, metastatic disease, etc.), treatments (dates, INN, route of administration, treatment protocols, reason for termination, etc.), and clinical events. Data is collected at each participating site by technicians who are specifically trained for the project using an electronic data collection (eDC) tool.

Data imported into the final database are controlled, recoded, and harmonized before import according to the data management plan. All coding procedures are predefined by the data manager. There is no transmission of individual data; all data are centralized within each center using a shared anonymous format. All data is exclusively obtained retrospectively; no attempts are made to recover non available data from the patient's medical record by contacting healthcare providers or patients.

ESME LC Data Platform aims to be a clinical and therapeutic database centralizing existing and available data from different sources used in the participating sites.

Data do not contain any personal data on patients. In compliance with the authorization delivered by the French Data Protection agency to Unicancer, only aggregated statistical reports and publication are released.

ELIGIBILITY:
Inclusion criteria :

* Adult (over 18)
* Treated (with radiotherapy or systemic anti-cancer treatment) for a lung cancer or diagnosed with metastatic lung cancer over the selection period at one of the participating site

Exclusion criteria

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients treated for lung cancer at one of the 38 French participating sites (Private comprehensive cancer centers and public hospitals).
Sampling Method: Non-Probability Sample
Enrollment: 70000 (Estimated)
Dates: Start 2017-10-02 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient characteristics | Baseline
  Age in years, Tobacco consumption, other exposures, Legal recognition as occupational disease, Medical history, History of other cancer, weight in kg and performance status (ECOG)
Tumor characteristics | Baseline
  Staging, Tumor size, sampling Method, histological type
Treatment patterns | From Baseline until 2024 (yearly basis)
  Drug, therapeutic class, treatment duration at each n treatment line

SECONDARY OUTCOMES:
Median overall survival | From date of diagnosis or first treatment until the date of death from any cause. Follow up until 2024
  Assessment of overall survival through treatment lines
Median surrogate endpoints for overall survival | From start date of the nth treatment line until the date of first applicable event. Follow up until 2024
  Surrogate endpoints (Progression-free Survival, Time to Progression, Time to Next Treatment) at each n treatment line.

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Laure Martin, Pharmacist, Study Director — UNICANCER
Locations (21):
- France (21):
  - Institut de Cancérologie de l'Ouest - Paul Papin, Angers
  - Institut Bergonié, Bordeaux
  - Centre François Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Hôpital Intercommunal de Créteil, Créteil
  - Centre Georges-François Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Institut Paoli-Calmettes, Marseille
  - Institut régional du Cancer Montpellier / Val d'Aurelle, Montpellier
  - Groupe Hospitalier Région Mulhouse et Sud Alsace - Hôpital Emile Muller, Mulhouse
  - Institut de cancérologie de l'Ouest - René Gauducheau, Nantes
  - Centre Antoine Lacassagne, Nice
  - Institut Curie, Paris
  - Institut Jean Godinot, Reims
  - Centre Henri Becquerel, Rouen
  - Institut Curie - Hôpital René Huguenin, Saint-Cloud
  - Centre Paul Strauss, Strasbourg
  - Institut Claudius Regaud, Toulouse
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Background] Robain M, Pérol M, Girard N, Debieuvre D, Coudert B, Madroszyk A, et al. Programme épidémio-stratégie médicoéconomique : une base nationale de données de vie réelle pour mieux comprendre la prise en charge du cancer bronchopulmonaire en France. Revue des Maladies Respiratoires. 2018 Jan;35:A106.
- [Result] Girard, N., M. Pérol, G. Simon, C. Audigier Valette, R. Gervais, D. Debieuvre, R. Schott, et al. " 90P - Real-world treatment patterns, clinical practice and outcomes for locally advanced, non resectable, non-small cell lung cancer from the French ESME Lung database ". Abstract Book of the European Lung Cancer Congress (ELCC) 10-13 April 2019, Geneva, Switzerland 30 (1 avril 2019): ii34. https://doi.org/10.1093/annonc/mdz067.006.
- [Result] Chouaid C, Filleron T, Debieuvre D, Perol M, Girard N, Dansin E, Lena H, Gervais R, Cousin S, Otto J, Schott R, Planchard D, Madroszyk A, Kaderbhai C, Dubray-Longeras P, Hiret S, Pichon E, Clement-Duchene C, Chenuc G, Simon G, Bosquet L, QUantin X. A Real-World Study of Patients with Advanced Non-squamous Non-small Cell Lung Cancer with EGFR Exon 20 Insertion: Clinical Characteristics and Outcomes. Target Oncol. 2021 Nov;16(6):801-811. doi: 10.1007/s11523-021-00848-9. Epub 2021 Oct 18. PMID 34661827
- [Result] Lamy T, Cabarrou B, Planchard D, Quantin X, Schneider S, Bringuier M, Besse B, Girard N, Chouaid C, Filleron T, Simon G, Baldini C. Biomarker Testing in Older Patients Treated for an Advanced or Metastatic Non-Squamous Non-Small-Cell Lung Cancer: The French ESME Real-Life Multicenter Cohort Experience. Cancers (Basel). 2021 Dec 24;14(1):92. doi: 10.3390/cancers14010092. PMID 35008257
- [Result] Griesinger F, Perol M, Girard N, Durand-Zaleski I, Zacharias S, Bosquet L, Janicke M, Quantin X, Groth A, Fleitz A, Calleja A, Patel S, Lacoin L, Daumont MJ, Penrod JR, Carroll R, Waldenberger D, Reynaud D, Thomas M, Chouaid C. Impact of immune checkpoint inhibitors on the management of locally advanced or metastatic non-small cell lung cancer in real-life practice in patients initiating treatment between 2015 and 2018 in France and Germany. Lung Cancer. 2022 Oct;172:65-74. doi: 10.1016/j.lungcan.2022.08.001. Epub 2022 Aug 6. PMID 36007281
- [Result] Chouaid C, Thomas M, Debieuvre D, Durand-Zaleski I, Zacharias S, Bosquet L, Groth A, Fleitz A, Calleja A, Patel S, Lacoin L, Daumont MJ, Penrod JR, Carroll R, Waldenberger D, Cotte FE, Audigier-Valette C, Griesinger F. Effectiveness of Nivolumab in Second-Line and Later in Patients with Advanced Non-Small Cell Lung Cancer in Real-Life Practice in France and Germany: Analysis of the ESME-AMLC and CRISP Cohorts. Cancers (Basel). 2022 Dec 13;14(24):6148. doi: 10.3390/cancers14246148. PMID 36551632
- [Result] Bringuier M, Carton M, Debieuvre D, Pasquier D, Perol M, Filleron T, Lena H, Quantin X, Simon G, Baldini C. Enrolment of older adults with advanced or metastatic non-small cell lung cancer in first-line clinical trials in the multicentre ESME cohort. J Geriatr Oncol. 2023 Mar;14(2):101423. doi: 10.1016/j.jgo.2022.101423. Epub 2023 Jan 17. PMID 36657245
- [Result] Chouaid C, Bosquet L, Girard N, Kron A, Scheffler M, Griesinger F, Sebastian M, Trigo J, Viteri S, Knott C, Rodrigues B, Rahhali N, Cabrieto J, Diels J, Perualila NJ, Schioppa CA, Sermon J, Toueg R, Erdmann N, Mielke J, Nematian-Samani M, Martin-Fernandez C, Pfaira I, Li T, Mahadevia P, Wolf J. An Adjusted Treatment Comparison Comparing Amivantamab Versus Real-World Clinical Practice in Europe and the United States for Patients with Advanced Non-Small Cell Lung Cancer with Activating Epidermal Growth Factor Receptor Exon 20 Insertion Mutations. Adv Ther. 2023 Mar;40(3):1187-1203. doi: 10.1007/s12325-022-02408-7. Epub 2023 Jan 18. PMID 36652175
- [Result] Belaroussi Y, Bouteiller F, Bellera C, Pasquier D, Perol M, Debieuvre D, Filleron T, Girard N, Schott R, Mathoulin-Pelissier S, Martin AL, Cousin S. Survival outcomes of patients with metastatic non-small cell lung cancer receiving chemotherapy or immunotherapy as first-line in a real-life setting. Sci Rep. 2023 Jun 13;13(1):9584. doi: 10.1038/s41598-023-36623-1. PMID 37311845
- [Result] Valette CA, Filleron T, Debieuvre D, Lena H, Perol M, Chouaid C, Simon G, Quantin X, Girard N. Treatment patterns and clinical outcomes of extensive stage small cell lung cancer (SCLC) in the real-world evidence ESME cohort before the era of immunotherapy. Respir Med Res. 2023 Nov;84:101012. doi: 10.1016/j.resmer.2023.101012. Epub 2023 Mar 27. PMID 37307617
- [Result] Heudel PE, de Montfort A, Debieuvre D, Chouaid C, Carton M, Audigier-Valette C, Filleron T, Chabaud S, Stancu A, Quantin X, Hiret S, Bosquet L, Blay JY. Reduced risk of secondary primary extra pulmonary cancer in advanced/metastatic lung cancer patients treated with immune checkpoint inhibitors. Lung Cancer. 2023 Aug;182:107280. doi: 10.1016/j.lungcan.2023.107280. Epub 2023 Jun 16. PMID 37339550
- [Result] Thomas QD, Quantin X, Lemercier P, Chouaid C, Schneider S, Filleron T, Remon-Masip J, Perol M, Debieuvre D, Audigier-Valette C, Justeau G, Loeb A, Hiret S, Clement-Duchene C, Dansin E, Stancu A, Pichon E, Bosquet L, Girard N, Du Rusquec P. Clinical characteristic and survival outcomes of patients with advanced NSCLC according to KRAS mutational status in the French real-life ESME cohort. ESMO Open. 2024 Jun;9(6):103473. doi: 10.1016/j.esmoop.2024.103473. Epub 2024 Jun 3. PMID 38833966
- [Result] Cabart M, Mourey L, Pasquier D, Schneider S, Lena H, Girard N, Chouaid C, Schott R, Hiret S, Debieuvre D, Quantin X, Madroszyk A, Dubray-Longeras P, Pichon E, Baranzelli A, Justeau G, Perol M, Bosquet L, Cabarrou B. Real-world overview of therapeutic strategies and prognosis of older patients with advanced or metastatic non-small cell lung cancer from the ESME database. J Geriatr Oncol. 2024 Sep;15(7):101819. doi: 10.1016/j.jgo.2024.101819. Epub 2024 Jul 26. PMID 39068144
- [Result] Thomas QD, Girard N, Bosquet L, Cavaillon S, Filleron T, Eltaief S, Chouaid C, Lena H, Debieuvre D, Perol M, Quantin X. Optimizing Treatment Strategies for Egfr-Mutated Non-Small-Cell Lung Cancer Treated with Osimertinib: Real-World Outcomes and Insights. Cancers (Basel). 2024 Oct 23;16(21):3563. doi: 10.3390/cancers16213563. PMID 39518004